CLINICAL TRIAL: NCT03310905
Title: Abdominal Wall Transplantation for the Reconstruction of Abdominal Wall Defects as Adjunct to Abdominal Solid Organ Transplantation
Brief Title: Abdominal Wall Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Linda Cendales, MD (Unknown); Kadiyala Ravindra, M.D. (Unknown); Detlev Erdmann, M.D. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00084054
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Transplant;Failure,Kidney; Transplant; Failure, Liver; Transplant; Failure, Bowel; Abdominal Wall Defect; Abdominal Wall Fistula; Abdominal Wall Hernia; Abdominal Wall Injury
Keywords: Research; Transplant; Abdominal Wall; Hernia
MeSH Terms: conditions — Hernia, Abdominal; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isolated Abdominal Wall Transplant (Experimental)
  Interventions: Procedure: Abdominal Wall Transplant alone
- Abdominal Wall with Solid Organ Transplant (Experimental)
  Interventions: Procedure: Abdominal Wall Transplant with another solid organ transplant

INTERVENTIONS:
Procedure: Abdominal Wall Transplant with another solid organ transplant — Transplant of abdominal wall in combination with another solid organ transplant.
  Arms: Abdominal Wall with Solid Organ Transplant
Procedure: Abdominal Wall Transplant alone — Abdominal Wall Transplant alone
  Arms: Isolated Abdominal Wall Transplant

SUMMARY:
The purpose of this protocol is to determine the safety and efficacy of abdominal wall transplantation as a treatment for the reconstruction of abdominal wall defects. Abdominal wall transplantation may be performed alone or in combination with another transplant.

DETAILED DESCRIPTION:
Within this protocol we propose to perform abdominal wall transplantation in 5 subjects, either as an isolated abdominal wall or in combination with another organ transplant. Each subject will be followed for a study period of 18 months.

Participants receiving an isolated abdominal wall or abdominal wall in combination with another organ transplant will receive the standard immunosuppression therapy as the non-vascularized composite allograft organ transplant. These patients will be studied to determine efficacy of the abdominal wall transplant to restore function of the defective abdominal wall for a study period of 18 months at Duke University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Candidates between 18-65 years old
* Willingness and legal ability to give consent
* Abdominal Wall in combination with another organ transplant: they must be eligible for the non-vascularized composite allograft organ transplant at Duke

Exclusion Criteria:

* Malignancy at evaluation or history of malignancy that precludes transplantation
* Pregnancy: Women who are of childbearing potential must have a negative serum pregnancy test within 48 hours of transplant and agree to use reliable contraception with two contraceptive methods for a minimum of 2 years following abdominal wall transplantation. Subjects seeking to become pregnant following 2 years will be made aware during the consent process that the effect of pregnancy on the transplanted abdominal wall and vice versa is unknown.
* Medical exclusion criteria for general anesthesia
* Ongoing substance abuse or history of untreated substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a viable abdominal wall transplant at 18 months | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda Cendales, MD, Principal Investigator — Duke University; Kadiyala Ravindra, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
At this time all data will be de-identified and there is no plan to make individual participant data available to other researchers.